CLINICAL TRIAL: NCT03872232
Title: A Randomized, Double-blind, Active-controlled, Multicenter Phase3 Trial to Evaluate the Efficacy and Safety of Co-administrated Rosuvastatin/Ezetimibe and Telmisartan in Patients With Primary Hypercholesterolemia and Essential Hypertension
Brief Title: Evaluating the Efficacy and Safety of Co-administrated Rosuvastatin/Ezetimibe and Telmisartan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROZETEL_RCT
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Hypercholesterolemia; Hypertension
MeSH Terms: conditions — Hypercholesterolemia; Hypertension | interventions — Ezetimibe; Rosuvastatin Calcium; Telmisartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ezetimibe/Rosuvastatin and Telmisartan (Experimental): 60 subjects will be assigned and the subjects will be administered "Ezetimibe/Rosuvastatin and Telmisartan" for 8 weeks.
  Interventions: Drug: Ezetimibe/Rosuvastatin; Drug: Telmisartan
- Ezetimibe/Rosuvastatin (Active Comparator): 60 subjects will be assigned and the subjects will be administered "Ezetimibe/Rosuvastatin" for 8 weeks.
  Interventions: Drug: Ezetimibe/Rosuvastatin
- Telmisartan (Active Comparator): 60 subjects will be assigned and the subjects will be administered "Telmisartan" for 8 weeks.
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Ezetimibe/Rosuvastatin — PO, Once daily(QD), 8weeks
  Other Names: Rosuvamibe Tab.
  Arms: Ezetimibe/Rosuvastatin; Ezetimibe/Rosuvastatin and Telmisartan
Drug: Telmisartan — PO, Once daily(QD), 8weeks
  Other Names: Micardis Tab.
  Arms: Ezetimibe/Rosuvastatin and Telmisartan; Telmisartan

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of co-administrated Rosuvastatin/Ezetimibe and Telmisartan in patients with primary hypercholesterolemia and essential hypertension.

DETAILED DESCRIPTION:
This trial is a phase 3 study to evaluate efficacy and safety of co-administrated Rosuvastatin/Ezetimibe and Telmisartan in patients with primary hypercholesterolemia and essential hypertension.

In "Rosuvastatin/Ezetimibe+Telmisartan" treatment group, 60 subjects will be assigned and the subjects administer "Rosuvastatin/Ezetimibe+Telmisartan" for 8 weeks.

In "Rosuvastatin/Ezetimibe" treatment group, 60 subjects will be assigned and the subjects administer "Rosuvastatin/Ezetimibe" for 8 weeks.

In "Telmisartan" treatment group, 60 subjects will be assigned and the subjects administer "Telmisartan" for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Subjects with hypertension and hyperlipidemia

Exclusion Criteria:

* Patient with known or suspected secondary hypertension
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Low density lipoprotein cholesterol (LDL-C) | Baseline, Week 8
  LDL-C change at Week 8 compared to Baseline
Mean sitting systolic blood pressure (MSSBP) | Baseline, Week 8
  MSSBP change at Week 8 compared to Baseline

SECONDARY OUTCOMES:
Mean sitting systolic blood pressure (MSSBP) | Baseline, Week 4
  MSSBP change at Week 4 compared to Baseline
Low density lipoprotein cholesterol (LDL-C) | Baseline, Week 4
  LDL-C change at Week 4 compared to Baseline
Mean sitting diastolic blood pressure (MSDBP) | Baseline, Week 4, Week 8
  MSDBP change at Week 4, 8 compared to Baseline
Total Cholesterol (TC) | Baseline, Week 4, Week 8
  TC change at Week 4, 8 compared to Baseline
High density lipoprotein cholesterol (HDL-C) | Baseline, Week 4, Week 8
  HDL-C change at Week 4, 8 compared to Baseline
Triglyceride (TG) | Baseline, Week 4, Week 8
  TG change at Week 4, 8 compared to Baseline
Low density lipoprotein cholesterol/High density lipoprotein cholesterol (LDL-C/HDL-C) | Baseline, Week 4, Week 8
  LDL-C/HDL-C change at Week 4, 8 compared to Baseline
Total Cholesterol/High density lipoprotein cholesterol (TC/HDL-C) | Baseline, Week 4, Week 8
  TC/HDL-C change at Week 4,8 compared to Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Soo Kim, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No